CLINICAL TRIAL: NCT05862116
Title: The Impact of Health Literacy on Quality of Life in Patients With Chronic Non-specific Low Back Pain: A Prospective Cohort Study
Brief Title: Impact of Health Literacy on Chronic Non-specific Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: CNSLBP1
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic non-specific low back pain: Patients with chronic non-specific low back pain.
  Interventions: Other: Survey form

INTERVENTIONS:
Other: Survey form — Patients will be asked to fill a survey form that consists of socio-demographic information, Turkish Health Literacy Scale -32, Short Form-36 Health Survey and Oswestry Disability Index.

SUMMARY:
This prospective cohort study aims to assess the impact of health literacy on the quality of life in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
This prospective cohort study will enroll patients with chronic non-specific low back pain. Patients will be assessed using Turkey Health Literacy Scale-32, Short Form-36 Health Survey, and Oswestry Disability Index. The correlation between health literacy and quality of life will be assessed with statistical tests.

ELIGIBILITY:
Inclusion Criteria:

-Chronic non-specific low back pain

Exclusion Criteria:

* Acute low back pain
* Radicular pain
* Spinal stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-specific low back pain that gave consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between health literacy and quality of life | 1 day
  Using the statistical analysis, this trial will assess the correlation between health literacy and quality of life. The Turkey Health Literacy Scale-32 results and Short Form-36 Health Survey results will be tested for possible correlation. Also, oswestry disability index and Turkey Health Literacy Scale-32 will also be tested for a possible correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request by the corresponding author.